CLINICAL TRIAL: NCT06051045
Title: Observational Study to Evaluate Efficacy, Safety and Biomarkers of Bulevirtide Treatment in Patients With Chronic Hepatitis D
Brief Title: Study to Evaluate Efficacy, Safety and Biomarkers of Bulevirtide Treatment in Chronic Hepatitis D Patients
Acronym: SEE-D
Status: Recruiting | Type: Observational
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Soo Aleman, Professor, MD, PhD, Karolinska University Hospital
Other Study IDs: SEE-D
Record Dates: First submitted 2023-09-06; First posted 2023-09-22 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Chronic Hepatitis D
MeSH Terms: conditions — Hepatitis D, Chronic | interventions — bulevirtide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biological sampling of blood, saliva and fecal samples and liver tissue (liver biopsy or fine needle aspiration
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Bulevirtide — Hepcludex, 2 mg daily subcutaneous injection

SUMMARY:
The aim is to assess the efficacy and specific safety in an observational study of patients with Chronic hepatitis D (CHD) with prospective follow-up, with antiviral treatment of 2 mg Bulevirtide (BLV) +/- PEG-IFNα-2a and +/- NA given as part of the patient's routine medical care. Also, explorative endpoints of biomarkers in peripheral blood, saliva, fecal sample and/or intrahepatic markers/signatures, and quality of life outcomes will be assessed.

DETAILED DESCRIPTION:
Chronic hepatitis D (CHD) is considered to be the most severe form of hepatitis. It is a rare disease in European Union countries, with status of an orphan disease. Historically, only pegylated interferon alfa-2a (PEG-IFNα-2a) +/- nucleos(t)ide analogues (NA) have been used off-label for treatment of CHD, with insufficient virological response and frequent relapse. The first in class entry inhibitor for treatment of CHD, bulevirtide (BLV), product name Hepcludex) has received status of conditional marketing authorization by the European Medical Agency (EMA) in July 2020.

This conditional approval was based on two phase 2 studies, with limited sample sizes. A phase 3 clinical trial of 150 participants is ongoing.

Besides need of more efficacy and safety data, knowledge about immunological cellular response in BLV treated and identification of biomarkers for treatment response is needed. Observational studies with biological samplings are thus needed.

We aimed therefore to assess the efficacy and specific safety in an observational study with prospective follow-up, with antiviral treatment of 2 mg BLV +/- PEG-IFNα-2a and +/- NA given as part of the patient's routine medical care. Also, explorative endpoints of biomarkers in peripheral blood, saliva, fecal sample and/or intrahepatic markers/signatures, and quality of life outcomes will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Diagnosis of chronic HBV/HDV co-infection.
3. Have compensated liver disease (presence of portal hypertension without ongoing hepatic decompensation as ascites, variceal bleeding and hepatic encephalopathy allowed).
4. Have indication for treatment of BLV, or already treated with BLV.
5. For female* participants:

   1. Postmenopausal for at least one year, or
   2. Surgically sterile (total hysterectomy or bilateral oophorectomy, bilateral tubal ligation, staples, or another type of sterilization), or
   3. Abstinence from heterosexual intercourse throughout the treatment period, or
   4. Willingness to use highly effective contraception (double barrier method or barrier contraception in combination with hormonal or intrauterine contraceptive) throughout the treatment period and for 6 months after last dose of the drugs in the study.
6. Male participants must agree to use a highly effective contraception (double barrier method or barrier contraception in combination with hormonal or intrauterine contraceptive used by female partners) throughout the treatment period and for 6 months after last dose of the drugs in the study.
7. Participants who are willing to give written informed consent

Exclusion Criteria:

1. Any contra-indications to treatment with BLV, including any intolerance or hypersensitivity to the active ingredient or other components of BLV.
2. Pregnant or breast-feeding women.
3. Patients with predictable difficulties of follow-up according to the investigator.
4. Any other condition that, in the opinion of Investigator, precludes the patient from taking part in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males and females from the age of 18 diagnosed with chronic hepatitis D
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-09-27 (Actual); Primary Completion 2033-03 (Estimated); Study Completion 2033-03 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with virological response of Hepatitis D virus (HDV) RNA < Limit of Detection (LoD) at FU 12 months after End of Treatment (EOT). | Continuously, up to 12 months
  Measurement of virological response of HDV RNA < LoD

SECONDARY OUTCOMES:
Percentage of patients with virological response of HDV RNA < LoD | At Baseline, 1 and 3 months, every 3 months after treatment start up to 9 months after date of EOT.
  Percentage of patients with virological response of HDV RNA < LoD at at month 1, 3 and every 3 months after treatment start, and FU month 3, 6, and 9 after EOT.
Percentage of patients with Hepatitis B surface antigen (HBsAg) < LoD | At Baseline, 1 and 3 months, every 3 months after treatment start up to 12 months after date of EOT.
  Percentage of patients with HBsAg < LoD at month 1 and 3, and every 3 months after treatment start, and FU month 3, 6, 9 and 12 after EOT.
Change of HBsAg from baseline | From Baseline every 3 months until end of study.
  Change of HBsAg from baseline every 3 months during study period.
Percentage of patients with HDV RNA < LoD or HDV RNA reduction of at least 2 log10 compared to baseline | At Baseline, 1 and 3 months, every 3 months after treatment start up to 12 months after date of EOT.
  Percentage of patients with HDV RNA < LoD or HDV RNA reduction of at least 2 log10 compared to baseline, at month 1 and 3, and every 3 months after treatment start, and FU month 3, 6, 9 and 12 after EOT.
Percentage of patients with virological relapse, defined as HDV RNA < LoD at EOT and increase of HDV RNA to > LoD after EOT | At 0, 3, 6, 9 and 12 months after date of EOT.
  Percentage of patients with virological relapse, defined as HDV RNA < LoD at EOT and increase of HDV RNA to > LoD after EOT, after EOT, at FU month 3, 6, 9 and 12 after EOT.
Percentage of patients with appearance of hepatitis B surface antibody (anti-HBs) | At 0, 3, 6, 9 and 12 months after date of EOT.
  Percentage of patients with appearance of hepatitis B surface antibody (anti-HBs) at EOT, and FU month 3, 6, 9 and 12 after EOT.
Percentage of patients with HBV DNA level < LoD | From Baseline every 3 months until end of study.
  Percentage of patients with HBV DNA level < LoD every 3 months during study period.
Percentage of patients with biochemical response, defined as normalization of alanine transaminase (ALT) | At Baseline, 1 and 3 months, every 3 months up to 12 months after date of EOT.
  Percentage of patients with biochemical response, defined as normalization of alanine transaminase (ALT), at month 1, 3 and every 3 months during treatment, and FU month 3, 6, 9 and 12 after EOT.
Percentage of patients with combined response, defined as HDV RNA < LoD or HDV RNA reduction of at least 2 log10 compared to baseline and Alanine Aminotransferase (ALT) normalization | At Baseline, at 1, 2 and 3 months, every 3 months up to 12 months after date of EOT.
  Percentage of patients with combined response, defined as HDV RNA < LoD or HDV RNA reduction of at least 2 log10 compared to baseline and ALT normalization, at month 1, 2 and 3, and every 3 months after treatment start, and FU month 3, 6, 9 and 12 after EOT.
Change of liver elasticity measurement level and percentage of AE of special interest | At Baseline, every 6 months until 12 months after date of EOT.
  Change of liver elasticity measurement level from baseline compared to the level at every 6 months during on-treatment, EOT, and FU month 6 and 12 after EOT.
  Percentage of AE of special interest: 1. Liver-related event, defined as new diagnoses of liver cirrhosis, HCC, or hepatic decompensation (ascites, variceal bleeding or hepatic encephalopathy); 2. Event of ≥ grade 3 hematological AE (in IFN treated); 3. Event of thyroid disorder (in IFN treated); 4. Event of injection site reaction; 5. Event of≥ grade 3 ALT increase.
Percentage of missed BLV doses during treatment | Continuously during treatment period until date of EOT.
  Percentage of missed BLV doses during treatment.
Percentage of patients with early discontinuation of treatment | Continuously during treatment period until date of EOT.
  Percentage of patients with early discontinuation of treatment and the reasons.
Serious Adverse Events | Continuously during study period until end of study.
  Percentage of patients with SAE.

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska University Hospital, Department of Infectious Diseases, Stockholm, Sweden